CLINICAL TRIAL: NCT00937820
Title: YM150 Long Term Study - Long-term Study in Patients With a History of Venous Thromboembolism
Brief Title: Prevention of Recurrence of Venous Thromboembolism in Patients With a History of Venous Thromboembolism
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Director, Astellas Pharma, Inc
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 150-CL-104
Record Dates: First submitted 2009-07-09; First posted 2009-07-13 (Estimated); Last update posted 2011-01-06 (Estimated); Status verified 2011-01

CONDITIONS: Venous Thromboembolism
Keywords: YM150; Bleeding; VTE; FXa inhibitor; Venous thromboembolism
MeSH Terms: conditions — Venous Thromboembolism; Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- YM150 group (Experimental)
  Interventions: Drug: YM150

INTERVENTIONS:
Drug: YM150 — oral

SUMMARY:
The study objective is to evaluate the efficacy and safety of oral YM150 for 52 weeks in patients with a history of venous thromboembolism.

ELIGIBILITY:
Inclusion Criteria:

* Subject has symptomatic VTE and/or asymptomatic deep vein thrombosis
* Written informed consent obtained before screening

Exclusion Criteria:

* Subject has history of deep vein thrombosis and/or pulmonary embolism
* Subject has a hemorrhagic disorder and/or coagulation disorder
* Subject has had clinically important bleeding occurred within 90 days prior to the screening visit
* Subject has an acute bacterial endocarditis
* Subject has uncontrolled severe or moderate hypertension, retinopathy, myocardial infarction or stroke
* Subject is receiving anticoagulants/antiplatelet agents
* Subject has a body weight less than 40 kg

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2009-06; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Joint incidence of deep vein thromboembolism or pulmonary thromboembolism | 52 weeks

SECONDARY OUTCOMES:
Incidence of each thromboembolism | 52 weeks
All cause mortality | 52 weeks
Incidence of bleeding event | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (5):
- Japan (5):
  - Chugoku
  - Chūbu
  - Kansai
  - Kantou
  - Tōhoku